CLINICAL TRIAL: NCT01204502
Title: Phase I/II Clinical Trial of T-cell Suicide Gene Therapy Following Haploidentical Stem Cell Transplantation
Brief Title: Suicide Gene Therapy Trial
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Changes in the clinical practice
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Biren Patel, Great Ormond Street Hospital for Children NHS Trust
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06MI04
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Haploidentical Stem Cell Transplantation
Keywords: Gene therapy; Haploidentical; Bone marrow transplant; Graft versus host disease; haploidentical stem cell transplantation; T-cell suicide gene therapy
MeSH Terms: conditions — Graft vs Host Disease

ARMS (1):
- HSVTK retrovirally-transduced donor T lymphocytes (Experimental): HSVTK retrovirally-transduced donor T lymphocytes will be given at 1 month intervals, providing that there is no significant GVHD
  * dose 1 5x104 cells/kg
  * dose 2 5x105 cells/kg
  Interventions: Biological: HSVTK retrovirally-transduced donor T lymphocytes

INTERVENTIONS:
Biological: HSVTK retrovirally-transduced donor T lymphocytes — HSVTK retrovirally-transduced donor T lymphocytes will be given at 1 month intervals, providing that there is no significant GVHD
  * dose 1 5x104 cells/kg
  * dose 2 5x105 cells/kg

SUMMARY:
Bone marrow or blood stem cell transplantation is used to treat a wide range of life-threatening conditions. T lymphocytes carried in the graft have powerful beneficial effects and play a vital role in the eradication of leukaemia and in fighting infection, but can also damage healthy tissues and cause graft-versus-host disease (GVHD).

To safeguard against GVHD, the investigators propose modifying T cells to encode a 'switch' so that they can be eliminated if problems arise.

Children receiving half-matched (haploidentical) transplants from a parent are most likely to benefit from this strategy. At present these patients receive blood stem cells from a parent, but the T cells are removed because the risk of serious GVHD is unacceptable. This means that they are much more likely to suffer from life threatening infections or experience a relapse of leukaemia. The investigators want to use gene therapy to produce "safe" T cells which can be used to strengthen the transplant and prevent these serious complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary immunodeficiencies, haematological malignancies or metabolic disorders at GOSH (children of both sexes, aged 0 to 16 years) undergoing haploidentical transplant
2. Both patient and donor must give informed consent in writing.
3. The donor must be willing, able and available for donation of T cells by collection of whole blood or leukapheresis.
4. The patient should be free of serious intercurrent illness.

Exclusion Criteria:

1. Donor unfit or unavailable
2. Donor positive for Hepatitis B or C, or HTLV-1, or HIV
3. Patient receiving Ganciclovir, Aciclovir, Cidofovir a result of active CMV, adenovirus, varicella zoster or herpes simplex infection infection
4. GVHD ≥ grade II before infusion of gene modified T cells
5. Serious intercurrent illness

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
T-cell reconstitution (as defined by CD4+ cells >300/mm3 & CD3+ cells >500/mm3) | 12 months after final dose
  T-cell reconstitution is measured until 12 months after administration of the final dose of gene modified cells

SECONDARY OUTCOMES:
Incidence of GvHD | 12 months after final dose
  Incidence of GvHD is measured until 12 months after administration of the final dose of gene modified cells
Patient survival | 12 months after final dose
  Patient survial is measured until 12 months after administration of the final dose of gene modified cells

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital for Children NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Qasim W, Gaspar HB, Thrasher AJ. T cell suicide gene therapy to aid haematopoietic stem cell transplantation. Curr Gene Ther. 2005 Feb;5(1):121-32. doi: 10.2174/1566523052997497. PMID 15638716
- [Derived] Zhan H, Gilmour K, Chan L, Farzaneh F, McNicol AM, Xu JH, Adams S, Fehse B, Veys P, Thrasher A, Gaspar H, Qasim W. Production and first-in-man use of T cells engineered to express a HSVTK-CD34 sort-suicide gene. PLoS One. 2013 Oct 21;8(10):e77106. doi: 10.1371/journal.pone.0077106. eCollection 2013. PMID 24204746